CLINICAL TRIAL: NCT07038980
Title: Investigation of the Effect of Smartphone Addiction on Neck Pain and the Structural and Mechanical Properties of Neck Muscles in Young Adults
Brief Title: Smartphone Addiction and Cervical Muscular Health
Status: Recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, ESRA PEHLIVAN, PhD, Saglik Bilimleri Universitesi
Other Study IDs: Smartphone Addiction&Neck
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Smartphone Addiction; Neck Pain
MeSH Terms: conditions — Internet Addiction Disorder; Neck Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Smartphone Addiction Group: Participants scoring above the cutoff values on the Smartphone Addiction Scale - Short Form (≥31 for males, ≥33 for females).
  Interventions: Other: Observational Assessment
- Non-Addicted Group: Participants who do not meet the addiction criteria according to the SAS-SF. These individuals demonstrate regular or low smartphone use and serve as a comparative control group for musculoskeletal outcomes.
  Interventions: Other: Observational Assessment

INTERVENTIONS:
Other: Observational Assessment — Participants in both groups undergo a one-time diagnostic evaluation consisting of:
  Smartphone Addiction Scale - Short Form (SAS-SF)
  Neck Disability Index (NDI)
  MyotonPRO measurement of cervical muscle tone, stiffness, and elasticity
  Pressure pain threshold measurement using a handheld algometer
  Social Media Addiction Scale (SMAS)
  No therapeutic or behavioral intervention is applied. All procedures are non-invasive and conducted for observational purposes only.

SUMMARY:
This cross-sectional observational study investigates how smartphone addiction affects neck pain severity, pressure pain threshold, and mechanical properties of cervical muscles in healthy young adults. Two groups-those with and without smartphone addiction-are compared based on validated addiction scales and objective muscle assessments using MyotonPRO and algometry.

DETAILED DESCRIPTION:
Smartphone addiction has become increasingly prevalent among young adults, often accompanied by poor posture and musculoskeletal complaints. This study aims to identify the differences in neck-related pain, disability, and mechanical muscle characteristics between addicted and non-addicted individuals. Participants are assessed using the Smartphone Addiction Scale - Short Form (SAS-SF), Social Media Addiction Scale (SMAS), Neck Disability Index (NDI), MyotonPRO for muscle tone/stiffness/elastance, and pressure algometry. The findings may contribute to the development of ergonomic and behavioral strategies for musculoskeletal health preservation in digital device users.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-30 years
* Actively using a smartphone
* Volunteer consent provided

Exclusion Criteria:

* Any diagnosed cervical spine pathology
* Neurological, rheumatological, or psychiatric disease
* Previous cervical surgery
* Lack of cooperation or inability to understand instructions

Ages: 18 Years to 30 Years | Sex: All
Age Groups: Adult
Study Population: The study population consists of healthy young adults aged between 18 and 30 years who are active smartphone users. All participants were university students without any known neurological, rheumatological, psychiatric, or musculoskeletal disorders affecting the cervical region. Individuals were classified into two groups based on their scores on the Smartphone Addiction Scale - Short Form (SAS-SF): smartphone-addicted and non-addicted. The population was chosen due to the increasing prevalence of smartphone use and associated postural complaints in this age group.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Quantitative Muscle Mechanical Assessment | Baseline
  A handheld digital palpation device used to measure biomechanical properties of superficial cervical muscles (tone, stiffness, elasticity). Measurements are taken bilaterally from specific muscles (e.g., platysma, SCM, upper trapezius, suboccipital muscles) in a resting position.

SECONDARY OUTCOMES:
Neck Disability Index (NDI) | Baseline
  A 10-item scale assessing the functional impact of neck pain on daily life, including activities such as driving, reading, work, sleep, and concentration. Each item is scored from 0-5; total scores reflect the severity of neck-related disability.
Smartphone Addiction Scale - Short Form (SAS-SF) | Baseline
  A 10-item, 6-point Likert-type scale used to classify participants as smartphone addicted or not. Validated cutoff values (≥31 for males, ≥33 for females) were used. This tool is used for group classification.
Social Media Addiction Scale (SMAS) | Baseline
  A 41-item, 5-point Likert scale evaluating participants' social media usage across four domains: preoccupation, emotional regulation, repetition, and conflict. It helps quantify social media behavior and its relation to neck dysfunction.
Pressure Algometry | Baseline
  Pressure pain thresholds were measured using a handheld algometer on bilateral cervical muscles. Participants were instructed to indicate when pressure became painful. Each site was measured three times, and the mean was recorded. Values reflect tissue sensitivity.

CONTACTS AND LOCATIONS:
Locations (1):
- Saglik Bilimleri Universitesi, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided